CLINICAL TRIAL: NCT04720144
Title: Multicenter Case-control Study of Breakthrough Invasive Mold Infections Under Posaconazole Prophylaxis
Brief Title: Breakthrough Invasive Mold Infections Under Posaconazole Prophylaxis (BIMI)
Acronym: BIMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Frederic Lamoth, Principal investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2020-01719
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Invasive Mold Infections; Breakthrough Invasive Mold Infections; Hematologic Malignancy; Hematologic Diseases
Keywords: Posaconazole; Antifungal prophylaxis
MeSH Terms: conditions — Hematologic Neoplasms; Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- bIMI cases: Adult (≥ 18 years old) patients with a hematologic malignancy receiving posaconazole prophylaxis (oral tablets or IV administration) for:
  i) Induction, consolidation or re-induction chemotherapy for acute leukemia or myelodysplastic syndrome (i.e. expected duration of neutropenia post-chemotherapy of ≥ 10 days) OR ii) Allogeneic hematopoietic stem cell transplant recipients during the post-transplantation phase (100-day post-transplantation) or later in case of intensified immunosuppression for moderate to severe graft vs host disease (GVHD).
  AND
  iii) Being diagnosed with proven or probable bIMI according to the EORTC-MSGERC classification (10) while on continuous posaconazole prophylaxis for at least 7 days.
- Controls: For each bIMI case, we will include 2 control cases fulfilling the following criteria:
  i) Receiving continuous posaconazole prophylaxis for at least 7 days
  ii) No diagnosis of proven, probable or possible IMI according to EORTC-MSGERC classification (10) during the entire hospital stay

SUMMARY:
Invasive mold infections (IMI) mainly affect patients with hematologic malignancies receiving intensive chemotherapy or after hematopoietic stem cell transplantation (HSCT). Prolonged neutropenia after remission induction chemotherapy (>10 days duration) and continuous immunosuppression in the context of prevention or therapy of graft versus host disease (GVHD) for HSCT recipients (first 100 days post-transplantation and thereafter if GVHD is present) are considered as periods at high risk of IMI.

Posaconazole prophylaxis is prescribed according to current guidelines to reduce the occurrence of IMI. Nevertheless, breakthrough IMI (bIMI), i.e. IMI occurring under mold-active prophylaxis, are still observed.

The investigators hypothesized that the epidemiology of bIMI (under posaconazole prophylaxis) differs from that of IMI occurring in the absence of mold-active antifungal prophylaxis. Because bIMI are rare events since the introduction of posaconazole prophylaxis, epidemiological data of bIMI are scarce.

This study aims to i) describe the epidemiology, clinical features, treatment and outcome of bIMI, ii) assess the causes of bIMI, iii) determine potential risk factors associated with the developllement of bIMI iv) assess the impact of bIMI on overall mortality.

Design

Retrospective and prospective, observational, case-control, multicenter, international study.

The retrospective part will enroll previously identified bIMI cases and control cases (1:2) over the last five years: October 1st 2015 to September 30st 2020.

The prospective part will enroll bIMI cases and control cases (1:2) occurring over a two-year period: October 1st 2020 to September 30st 2022.

Setting

The aim is to enroll 10 to 15 European centers with dedicated units for hematologic cancer patients. Currently, six centers have confirmed their participation (from Switzerland and Germany).

Study Population

Adult (≥ 18 years old) patients with a hematologic malignancy receiving posaconazole prophylaxis during induction, consolidation or re-induction chemotherapy or after HSCT.

Cases : patients receiving posaconazole prophylaxis for at least 7 days and diagnosed with bIMI proven or probable according to EORTC-MSGERC.

Controls: patients receiving posaconazole prophylaxis for at least 7 days, without diagnosis of bIMI possible, probable or proven according to EORTC-MSGERC.

The objective is to enroll about 100 bIMI cases and 200 controls.

ELIGIBILITY:
Inclusion Criteria:

* Cases:

Adult (≥ 18 years old) patients with a hematologic malignancy receiving posaconazole prophylaxis (oral tablets or IV administration) for:

i) Induction, consolidation or re-induction chemotherapy for acute leukemia or myelodysplastic syndrome (i.e. expected duration of neutropenia post-chemotherapy of ≥ 10 days)

OR

ii) Allogeneic hematopoietic stem cell transplant recipients during the post-transplantation phase (100-day post-transplantation) or later in case of intensified immunosuppression for moderate to severe graft vs host disease (GVHD).

AND

iii) Being diagnosed with proven or probable bIMI according to the EORTC-MSG classification (10) while on continuous posaconazole prophylaxis for at least 7 days.

* Controls:

For each bIMI case, we will include 2 control cases fulfilling the following criteria:

i) Receiving continuous posaconazole prophylaxis for at least 7 days

ii) No diagnosis of proven, probable or possible IMI according to EORTC-MSG classification (10) during the entire hospital stay.

And matched to bIMI cases according to the following criteria:

iii) Hospitalization in the same ward within the same year (+/- 12 months interval)

iv) Same underlying condition related to hematologc cancer: a) HSCT within 100 days post-engraftment, b) HSCT > 100 days post-engraftment with intensified immunosuppressive regimen for severe GVHD, c) induction chemotherapy for acute myeloid or lymphoid leukemia, or myelodysplastic syndrome, d) other hematologic disorders (e.g. aplastic anemia) with prolonged neutropenia and/or immunosuppressive regimen.

Exclusion Criteria:

* Patients with a diagnosis of possible IMI according to the EORTC-MSG classification.
* Patients with a positive fungal biomarker in serum (e.g. galactomannan or beta-glucan) in the absence of clinical or radiological criteria of IMI according to the EORTC-MSG classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with hematologic malignancies under posaconazole prophylaxis for one of the above mentionned reasons.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Epidemiological description of bIMI | At inclusion
  * Assessment of the cause of bIMI (intrinsically resistant mold pathogen vs susceptible mold pathogen but insufficient posaconazole serum concentration vs unknown)
  * Description of clinical features, treatment and outcome of bIMI
Assessment of the risk factors of bIMI | At inclusion
  • Univariate and multivariate analyses of the parameters associated with an increased risk of bIMI (in particular, the association of a threshold of posaconazole concentration and bIMI) by comparison of bIMI cases with controls (posaconazole prophylaxis and no bIMI)

SECONDARY OUTCOMES:
Assessment of the impact of bIMI on overall mortality | 6 weeks and 12 weeks after inclusion
  • Comparison of mortality rate (6 and 12 weeks) between bIMI and control cases.
Assessment of factors influencing outcomes of bIMI | 6 weeks and 12 weeks after inclusion
  • Univariate and multivariate analysis of predictors of mortality (6 and 12 weeks) among bIMI cases.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Lamoth, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (8):
- Medical University of Innsbruck, Innsbruck, Austria
- University Hospital Cologne, Cologne, Germany
- Switzerland (6):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Hôpital Cantonal de Fribourg, Fribourg
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Kantonsspital St.Gallen, Sankt Gallen